CLINICAL TRIAL: NCT04034940
Title: Correlations Between Oxidative Stress Biomarkers, h-FABP and Left Ventricular Dysfunction in Patients With Acute Myocardial Infarction Undergoing Primary PCI
Acronym: OxiSTEMIhFABP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Grigore T. Popa University of Medicine and Pharmacy (Other)
Collaborators: Cardiovascular Diseases Institute IASI, Romania (Unknown)
Responsible Party: Principal Investigator, Professor Adrian Covic, Professor, Vice-rector, Grigore T. Popa University of Medicine and Pharmacy
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: OxiSTEMI01
Record Dates: First submitted 2019-07-24; First posted 2019-07-29 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: STEMI; Oxidative Stress; Oxidative Stress Induction; Primary PCI; hFABP; Left Ventricular Dysfunction; BCM
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Ventricular Dysfunction, Left | interventions — Fatty Acid Binding Protein 3

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- primary PCI STEMI patients (Other): All Patients with AMI refered for primary PCI in single center
  Interventions: Other: Dosing Oxidative stress biomarkers & hFABP in STEMI pPCI patients

INTERVENTIONS:
Other: Dosing Oxidative stress biomarkers & hFABP in STEMI pPCI patients — Dosing oxidative stress biomarkers and hFABP in STEMI pPCI

SUMMARY:
The investigators intend to evaluate Oxidative Stress biomarkers through a. Catalase Activity Assay; b. Lipid Peroxidation Assay; c. SOD Assay; d. Total Antioxidant Capacity Assay; e. Glutathione Peroxidase at patients with acute myocardial infarction STEMI referred for primary PCI; The investigators also aim to evaluate cardiac necrosis by measuring Heart Fatty Acid Binding Protein (H-FABP), TnI, CK, CK-MB, LDH and AST in these patients with acute myocardial infarction referred for primary PCI; Also, the investigators intend to evaluate body composition through bioimpedance spectroscopy (BCM - Fresenius Care) at the moment of admission.

The investigators aim to fully characterise these patients through oxidative millieu, hFABP and make correlations with LVEF dysfunction.

DETAILED DESCRIPTION:
Gathered data:

* Descriptive general demographic data;
* Previous pathologies (ischemic heart disease, peripheral arterial disease, stroke, heart failure, previous percutaneous coronary interventions, coronary artery bypass grafting - CABG, known renal disease);
* Cardiovascular risk factors (age, weight, height, abdominal perimeter, body mass index, smoking, sedentariness, diabetes, hypertension, dyslipidaemia);
* Oxidative Stress biomarkers: Catalase Activity Assay; Lipid Peroxidation Assay; SOD Assay; Total Antioxidant Capacity Assay; Glutathione ;
* Cardiac necrosis markers: Heart Fatty Acid Binding Protein (H-FABP), TnI, CK, CK-MB, LDH and OGT;
* Routine biological data;
* Metabolic data (obtained from two body composition monitoring evaluations - before and 12 hours after coronary intervention) - body water, body fat tissue;
* Information regarding primary PCI (less than 12 hours of ischemic symptoms);
* Coronarographic details, type of used stent, periprocedural specific complications, final TIMI - thrombolysis in myocardial infarction - flow);
* Echocardiography at admission (LVEF);
* Measurement of arterial stiffness through Sphigmocore pulsed-wave-velocity (24 hrs post-procedural, 2 velocities: carotid - femoral and carotid - radial);
* Calculating of cardiovascular risk scores: Syntax Score, Framingham score, ASSIGN score, QRISK2 score, PROCAM score, CRUSADE score, GRACE score, CHADS VASc score, MESA score, ASCVD score, Hamilton Depression Rating Scale (HAM-D), Hamilton Rating Scale for Anxiety;
* In-hospital and one month follow-up MACE.

ELIGIBILITY:
Inclusion Criteria:

* Adults with ST elevation Myocardial Infarction (<12h) diagnostic confirmed;
* Included in the Romanian National Programme of Primary Percutaneous Revascularisation (for who the Guidelines recommend primary PCI);

Exclusion Criteria:

* Patients who do not sign informed consent for primary PCI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-08 (Estimated); Primary Completion 2020-07 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Oxidative Stress status in Acute Myocardial Infarction Patients undergoing primary PCI | 1 year
  Assessment of oxidative stress status by measuring Catalase Activity Assay; Lipid Peroxidation Assay; SOD Assay; Total Antioxidant Capacity Assay; Glutathione Peroxidase.
2. Cardiac necrosis status in Acute Myocardial Infarction Patients undergoing primary PCI. | 1 year
  Assessment of cardiac necrosis by measuring Heart Fatty Acid Binding Protein (H-FABP), TnI, CK, CK-MB, LDH and AST

SECONDARY OUTCOMES:
Hydation Status in Acute Myocardial Infarction Patients undergoing primary PCI. | 1 year
  Assessment of hydration status through body composition monitoring BCM.

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Covic, Professor, Principal Investigator — University of Medicine and Pharmacy "Gr. T. Popa" Iasi, Romania
Locations (1):
- Cardiovascular Diseases Institute Iasi, Iași, Iaşi, Romania

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.